CLINICAL TRIAL: NCT05223192
Title: The Effects of Entrainment on Respiratory Stability and Cerebral Oxygenation in Preterm Infants
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Joanne Loewy, Associate Clinical Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY-21-01783
Record Dates: First submitted 2022-01-24; First posted 2022-02-03 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Prematurity
Keywords: music therapy; ocean disc; prematurity; vital signs; cerebral oxygenation
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Participants in this group will receive the ocean disc music therapy entrainment intervention
  Interventions: Behavioral: Music Therapy Entrainment with Ocean Disc Intervention
- Control group (No Intervention): Participants in this group will not receive any intervention

INTERVENTIONS:
Behavioral: Music Therapy Entrainment with Ocean Disc Intervention — The studied intervention regards live entrainment with the ocean disc. Entrainment involves the use of an external stimulus, in the case of this study, an ocean disc instrument. Motion of the disc creates sounds in synchrony with the breathing of the infant and then in turn can control and influence the infant's regulation of the breath.
  Arms: Intervention group

SUMMARY:
Infants born prematurely at will be asked to participate in this randomized controlled trial at a corrected gestational age of 24-37 weeks. Infants will be randomly selected to each of the two groups: intervention and control. Infants in the treatment group will receive six intervention days over a two-week period, 3 sessions per week. Each intervention day consists of each of the two interventions in a random sequence: no intervention/silence and live ocean disc instrument intervention. The sound decibel level will also be recorded and maintained at 40-65dB to prevent overstimulation. Each infant will thus receive control and ocean disc intervention on the same day in the NICU. Interventions will be given in a randomized order (i.e., first ocean disc or first silence, randomized to AM or PM), with observation occurring for 10 minutes before each intervention, 15 minutes during each intervention, and 10 minutes after each per session. There will be 3 sessions per week for a two-week randomized treatment schedule. For each infant, data on total apnea time, mean respiratory rate, heart rate, O2 levels and behavior rating during will be collected. The sound decibel level will also be recorded and maintained at 40-65dB to prevent overstimulation and hearing damage. Near-infrared light spectroscopy (NIRS) data on cerebral oxygenation will also be collected. Observations will be recorded on the infant's activity or when change occurs, such as a pacifier falling out. Parents and nurses will be asked to behave as they normally would during routine care.

ELIGIBILITY:
Inclusion Criteria:

* Newborns born at 24-37 weeks' gestation at Mount Sinai hospital
* Newborn is considered appropriate for clinically indicated music therapy

Exclusion Criteria:

* Infant not expected to survive 24 hours from the time of study entry (To be assessed by a member of the NICU Faculty other than the PI)
* Infant of uncertain viability (gestation <23 weeks, birth weight <500 grams)
* Known or suspected genetic disorder (e.g., Trisomy 21)
* Identified hearing disorder

Ages: 24 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 118 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Heart Rate | 14 days
Respiratory Rate | 14 days
Oxygen-Saturation Level | 14 days
Weight | 14 days
Cerebral oxygen saturation | 14 days
  Cerebral oxygen saturation measured using NIRS

CONTACTS AND LOCATIONS:
Overall Officials: Joanne V Loewy, DA, MT-BC, LCAT, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Hospitals, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
IPD will be made available upon reasonable request to corresponding author